CLINICAL TRIAL: NCT00943150
Title: A Prospective, Randomized, Controlled Two-arm Superiority Study to Evaluate Use of the PEAK PlasmaBlade™ 4.0 in Abdominoplasty
Brief Title: PEAK PlasmaBlade™ vs. Traditional Electrosurgery in Abdominoplasty
Acronym: PRECISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEAK VP-00055
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-11

CONDITIONS: Elastosis
Keywords: Abdominoplasty; PlasmaBlade; Electrosurgery; PEAK Surgical; Medtronic Advanced Energy; Medtronic
MeSH Terms: conditions — Hyperthermia | interventions — Standard of Care; Electrocoagulation; Electrosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEAK PlasmaBlade (Experimental): The PEAK PlasmaBlade will be used for the abdominoplasty procedure.
  Interventions: Device: PEAK PlasmaBlade
- Standard of Care (SOC) (Active Comparator): The scalpel and electrocautery will be used for the abdominoplasty procedure.
  Interventions: Procedure: Standard of Care (SOC)

INTERVENTIONS:
Device: PEAK PlasmaBlade — The PEAK PlasmaBlade will be used for the abdominoplasty procedure.
  Other Names: PlasmaBlade
  Arms: PEAK PlasmaBlade
Procedure: Standard of Care (SOC) — The scalpel and electrocautery will be used for the abdominoplasty procedure.
  Other Names: Bovie; electrocautery; electrosurgery
  Arms: Standard of Care (SOC)

SUMMARY:
The objective of this clinical study is to evaluate healing of incisions made with the PEAK PlasmaBlade 4.0 compared to scalpel and traditional electrosurgery (Bovie); to monitor and record key post-operative metrics following abdominoplasty with the PEAK PlasmaBlade 4.0 versus current standard of care (SOC); and to evaluate performance metrics of the PEAK PlasmaBlade 4.0 during abdominoplasty.

DETAILED DESCRIPTION:
Abdominoplasty is a cosmetic surgical procedure performed to correct abdominal elastosis with skin and fat redundancy. During the procedure, a scalpel and traditional electrosurgical device are used to cut away this excess skin and fat from the abdomen and the underlying muscles are tightened together with sutures.

The PEAK PlasmaBlade™ uses pulsed radiofrequency (RF) energy to enable precision cutting and coagulating at the point of application, without the thermal damage to surrounding tissues that is normally seen with traditional electrosurgery. The PlasmaBlade has received FDA clearance for use in plastic, general, and ear, nose, and throat (ENT) surgery, and has demonstrated significantly reduced serous drainage in tissue reduction surgeries, like abdominoplasty.

A total of twenty (20) human subjects were recruited from the local community against standardized inclusion/exclusion criteria. Once enrolled, each patient underwent placement of three sets of full-thickness comparison incisions in their abdominal skin with a standard scalpel, PlasmaBlade, and traditional electrosurgery at six (6) and three (3) weeks prior to abdominoplasty, and on the day of surgery under general anesthesia. Subjects were then randomized to undergo abdominoplasty with the PlasmaBlade or the SOC (scalpel and traditional electrosurgery). Following abdominoplasty, harvested healed incisions were submitted for histological analysis and burst strength testing and additional data were recorded in the 10 day post-operative period.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 60 years old
2. Physically healthy, stable weight, non-smoker
3. Protruding abdomen, excess fat and skin and/or weak abdominal muscles qualifying for abdominoplasty.
4. Subject must understand the nature of the procedure and provide written informed consent prior to the procedure.
5. Subject must be willing and able to comply with specified follow-up evaluations.
6. Female subjects must either be no longer capable of reproduction or taking acceptable measures to prevent pregnancy during the study, and have a negative pregnancy test prior to participation in the study.

Exclusion Criteria:

1. Age younger than 25 or greater than 60 years old
2. Anticoagulation therapy which cannot be discontinued
3. Smoking (any kind)
4. Diabetes (any type)
5. Infection (local or systemic)
6. Cognitive impairment or mental illness
7. Severe cardiopulmonary deficiencies
8. Known coagulopathy
9. Immunocompromised
10. Kidney disease (any type)
11. Subjects who are pregnant or lactating
12. Currently taking any medication known to affect healing
13. Subjects who are status-post gastric banding or gastric bypass
14. Reproductive age females who will not take acceptable measures to prevent pregnancy during the study.
15. Recent history of abdominal surgery or prior abdominoplasty.
16. Subjects who are known to be HIV or Hepatitis (any) positive
17. Currently enrolled in another investigational device or drug trial
18. Unable to follow instructions or complete follow-up

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard L Rosenberg, MD, Principal Investigator — El Camino Hospital
Locations (1):
- El Camino Surgery Center, Mountain View, California, United States

REFERENCES:
- [Derived] Ruidiaz ME, Messmer D, Atmodjo DY, Vose JG, Huang EJ, Kummel AC, Rosenberg HL, Gurtner GC. Comparative healing of human cutaneous surgical incisions created by the PEAK PlasmaBlade, conventional electrosurgery, and a standard scalpel. Plast Reconstr Surg. 2011 Jul;128(1):104-111. doi: 10.1097/PRS.0b013e31821741ed. PMID 21701326

RESULTS

PARTICIPANT FLOW:
Groups:
- PEAK PlasmaBlade: The PEAK PlasmaBlade for the abdominoplasty procedure.
Period: Overall Study
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age Continuous [Mean (Full Range); unit: years] | 42.11 (9.41) [28 to 56] | 44.40 (10.72) [28 to 58] | 43.26 [28 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Acute Thermal Injury Depth
Description: Histological samples were created by first incising the area to be resected with all 3 modalities (PEAK PlasmaBlade, electrocautery, and scalpel) at 6 and 3 weeks before the operation. Then, the incised tissue was resected during the abdominoplasty and was assessed by analyzing incisions created in the resected area for histological measures.
  Acute thermal injury depth was assessed by incising the resected area during the abdominoplasty operation.
Time Frame: Immediately postoperative
Measure: Mean (Standard Deviation); unit: micrometers
Groups:
- PEAK PlasmaBlade: A surgical instrument that uses pulsed radiofrequency (RF) energy for the cutting and coagulation of soft tissue (skin and subcutaneous tissues) with the precision of a scalpel and hemostatic capability of traditional electrosurgery.
- Electrocautery: The standard of care for abdominoplasty consists of scalpel (for the skin incision) and traditional electrosurgery (for the subcutaneous dissection). Traditional electrosurgical instruments are used for the cutting and coagulation of soft tissues.
Arm/Group | PEAK PlasmaBlade | Electrocautery
Number analyzed (Participants) | 10 | 10
micrometers | 195 (127) | 763 (208)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Electrocautery; Test type: Superiority or Other; p < 0.001, Regression, Linear

2. Primary Outcome: Inflammatory Cell Count
Description: Histological samples were created by first incising the area to be resected with all 3 modalities (PEAK PlasmaBlade, electrocautery, and scalpel) at 6 and 3 weeks before the operation. Then, the incised tissue was resected during the abdominoplasty and was assessed by analyzing incisions created in the resected area for histological measures.
Time Frame: 0, 3, and 6 weeks
Measure: Mean (Standard Deviation); unit: cells per square millimeter
Groups:
- Electrosurgery; Scalpel: The standard of care for abdominoplasty consists of scalpel (for the skin incision) and traditional electrosurgery (for the subcutaneous dissection). Traditional electrosurgical instruments are used for the cutting and coagulation of soft tissues.
Arm/Group | PEAK PlasmaBlade | Electrosurgery | Scalpel
Number analyzed (Participants) | 20 | 20 | 20
cells per square millimeter
  CD3+ 0 weeks | 93 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 120 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 138 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable.
  CD3+ 3 weeks | 207 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 239 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 171 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable.
  CD3+ 6 weeks | 216 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 223 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 196 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable.
  CD68+ 0 weeks | 71 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 75 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 87 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable.
  CD68+ 3 weeks | 201 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 263 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 173 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable.
  CD68+ 6 weeks | 232 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 185 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable. | 202 (NA) — Study was conducted by PEAK Surgical before acquisition by Medtronic. The standard deviations for these outcome measures were not retrievable.
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Electrosurgery vs Scalpel; CD3+ at 0 weeks; Test type: Superiority or Other; p = 0.33, ANOVA
Statistical Analysis 2: Comparison: PEAK PlasmaBlade vs Electrosurgery vs Scalpel; CD3+ at 3 weeks; Test type: Superiority or Other; p = 0.02, ANOVA
Statistical Analysis 3: Comparison: PEAK PlasmaBlade vs Electrosurgery vs Scalpel; CD3+ at 6 weeks; Test type: Superiority or Other; p = 0.71, ANOVA
Statistical Analysis 4: Comparison: PEAK PlasmaBlade vs Electrosurgery vs Scalpel; CD68+ at 0 weeks; Test type: Superiority or Other; p = 0.67, ANOVA
Statistical Analysis 5: Comparison: PEAK PlasmaBlade vs Electrosurgery vs Scalpel; CD68+ at 3 weeks; Test type: Superiority or Other; p = 0.01, ANOVA
Statistical Analysis 6: Comparison: PEAK PlasmaBlade vs Electrosurgery vs Scalpel; CD68+ at 6 weeks; Test type: Superiority or Other; p = 0.48, ANOVA

3. Secondary Outcome: Total Drainage Output
Time Frame: 0 to 10 days postoperatively
Population: One subject was removed from the analysis of secondary variables owing to a protocol deviation.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 9 | 10
mL | 654.89 (217.74) | 887.70 (325.79)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Test type: Superiority or Other; p = 0.1128, Exact Wilcoxon rank-sum test

4. Secondary Outcome: Change in Hemoglobin
Description: The outcome measure is reported as change in hemoglobin, not the hemoglobin value itself.
Time Frame: Intraoperative
Population: One subject was removed from the analysis of secondary variables owing to a protocol deviation.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 9 | 10
g/dL | -0.68 (1.03) | -1.62 (1.21)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Test type: Superiority or Other; p = 0.0898, Exact Wilcoxon test

5. Secondary Outcome: Narcotic Consumption
Description: Narcotic medications were coded to Fentanyl microgram equivalent units per kilogram.
Time Frame: Intraoperative and postoperative (0 to 10 days)
Population: One subject was removed from the analysis of secondary variables owing to a protocol deviation.
Measure: Mean (Standard Deviation); unit: Fentanyl microgram units/g
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 9 | 10
Fentanyl microgram units/g
  Intraoperative | 3.82 (2.26) | 4.92 (1.72)
  Postoperative (0 to 10 days) | 2.39 (2.26) | 3.33 (2.75)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Intraoperative narcotic use comparison; Test type: Superiority or Other; p = 0.0760, Exact Wilcoxon test
Statistical Analysis 2: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Postoperative narcotic use comparison; Test type: Superiority or Other; p = 0.5900, Exact Wilcoxon test

6. Secondary Outcome: Postoperative Pain Levels
Description: Wong-Baker FACES Visual Analog Scale, 0 (no hurt) to 10 (hurts worst). The results represent the mean of each subject's mean pain scores over 10 days.
Time Frame: Postoperative (0 to 10 days)
Population: One subject was removed from the analysis of secondary variables owing to a protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 9 | 10
units on a scale | 2.15 (1.05) | 3.30 (2.72)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Test type: Superiority or Other; p = 0.4589, Exact Wilcoxon test

7. Secondary Outcome: Activity Level
Description: Sum of activity over 10 days postoperatively using a 0 (0% of normal) to 100 (100% of normal) visual analog scale. Subjects circled a number representing their activity level by tens (e.g., 10% of normal, 20% of normal). Subjects completed the scale daily through day 10. The results represent the mean cumulative value per patient.
Time Frame: Postoperative (0 to 10 days)
Population: One subject was removed from the analysis of secondary variables owing to a protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 9 | 10
units on a scale | 452.78 (139.57) | 347.00 (165.92)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Test type: Superiority or Other; p = 0.999, Exact Wilcoxon test

8. Secondary Outcome: Diet Volume
Description: Sum of diet volume (i.e., how much food the subject ate) over 10 days postoperatively using a 0 (0% of normal) to 100 (100% of normal) visual analog scale. Subjects circled a number representing their diet volume by tens (e.g., 10% of normal, 20% of normal). Subjects completed the scale daily through day 10. The results represent the mean cumulative value per patient.
Time Frame: Postoperative (0 to 10 days)
Population: One subject was removed from the analysis of secondary variables owing to a protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 9 | 10
units on a scale | 701.11 (160.97) | 470.50 (243.35)
Statistical Analysis 1: Comparison: PEAK PlasmaBlade vs Standard of Care (SOC); Test type: Superiority or Other; p = 0.0412, Exact Wilcoxon test

ADVERSE EVENTS:
Arm/Group | PEAK PlasmaBlade | Standard of Care (SOC)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEAK PlasmaBlade (N=10) | Standard of Care (SOC) (N=10)
Seroma (Surgical and medical procedures) | 0 (0) | 1 (1)
Extended drainage period (Surgical and medical procedures) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less